CLINICAL TRIAL: NCT05456308
Title: What is the Optimal Technique for Hydrodistention? First Prospective Study Evaluating the Effect of Pressure, Duration and Number of Hydrodistentions on Patients with Interstitial Cystitis
Brief Title: What is the Optimal Technique for Hydrodistention?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, James Clemens, Research Professor of Urology and Professor of Urology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00212141
Record Dates: First submitted 2022-07-05; First posted 2022-07-13 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
Keywords: Hydrodistension
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Intervention Model Description: Participants will be randomly selected to one of the arms described. There are three variables that they will be assigned: the pressure of fluid in the bladder that will be filled, the duration of time that the fluid will be held in the bladder, and the number of times the procedure is completed.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and statistician blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Pressure (30 centimeters), Duration (1 minute), Number of times done (1) (Experimental)
  Interventions: Procedure: Hydrodistention during cystoscope
- Pressure (30 centimeters), Duration (2 minute), Number of times done (1) (Experimental)
  Interventions: Procedure: Hydrodistention during cystoscope
- Pressure (30 centimeters), Duration (1 minute), Number of times done (2) (Experimental)
  Interventions: Procedure: Hydrodistention during cystoscope
- Pressure (80 centimeters), Duration (1 minute), Number of times done (1) (Experimental)
  Interventions: Procedure: Hydrodistention during cystoscope
- Pressure (80 centimeters), Duration (2 minute), Number of times done (1) (Experimental)
  Interventions: Procedure: Hydrodistention during cystoscope
- Pressure (80 centimeters), Duration (1 minute), Number of times done (2) (Experimental)
  Interventions: Procedure: Hydrodistention during cystoscope
- Pressure (30 centimeters), Duration (2 minute), Number of times done (2) (Experimental)
  Interventions: Procedure: Hydrodistention during cystoscope
- Pressure (80 centimeters), Duration (2 minute), Number of times done (2) (Experimental)
  Interventions: Procedure: Hydrodistention during cystoscope

INTERVENTIONS:
Procedure: Hydrodistention during cystoscope — Hydrodistention for treatment of interstitial cystitis will be performed. Participants will be randomly selected to one of the arms described. There are three variables that they will be assigned: the pressure of fluid in the bladder that will be filled, the duration of time that the fluid will be held in the bladder, and the number of times the procedure is completed.

SUMMARY:
This research study is being done to learn what is the best way to perform hydrodistention. Eligible participants will be enrolled and have follow-up for three months after surgery.

The study team hypothesizes that changes in hydrodistention technique, including pressure, number of distention, and duration of distention, leads to no or minimal changes in symptom improvement for patients with Interstitial cystitis/bladder pain syndrome (IC/BPS).

DETAILED DESCRIPTION:
Hydrodistention is a procedure designed to treat bladder and pelvic symptoms in patients with interstitial cystitis. A camera is placed inside the bladder and the bladder is filled with fluid. This procedure "resets" the signals between the bladder and brain, in order to reduce the symptoms of interstitial cystitis (such as bladder pain, urinary urgency/frequency/dysuria, incontinence, incomplete emptying, etc).

However, it is still unknown the best way to perform hydrodistention. Doctors do not know how much fluid to put in the bladder, how long to keep the fluid in the bladder, and how many times to fill the bladder.

ELIGIBILITY:
Inclusion Criteria:

* Patients with IC/BPS who have failed first/second line treatments (behavioral therapy, medications) for greater than 3 months
* Have not had hydrodistention performed in the past 3 months
* Have not had botox or Percutaneous tibial nerve stimulation (PTNS) performed in the past 3 months

Exclusion Criteria:

* Patients with known hunner's lesions
* Patients with interstim
* Patients with positive urinalysis/culture consistent with urinary tract infection (UTI)
* History of urethral, bladder, prostate, uterine, cervical, vaginal cancer
* History of augmentation cystoplasty or cystectomy
* History of urethral diverticulum, urethral stricture, pelvic radiation
* Patients with spinal cord injuries
* History of dementia, parkinson's disease, multiple sclerosis, spina bifida, paraplegia/quadriplegia, cerebral palsy, stroke
* Neurogenic bladder patients
* Anuric patients
* Tuberculous cystitis
* Cyclophosphamide treatment
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in the interstitial cystitis symptom index (ICSI) from baseline to 1-month | baseline to 1 month
  Identify the optimal technique for hydrodistention, including the optimal pressure (30 vs 80cc), number of hydrodistentions (one vs two), duration of each hydrodistention (one vs two minutes) as quantified by Changes in the interstitial cystitis symptom index (ICSI)f rom baseline to 1-month.
  The O'Leary-Sant questionnaire is composed of the Interstitial Cystitis Symptom Index (ICSI) and Problem Index (ICPI) which contains four questions related to urinary and pain symptoms. For the ICSI (score range: 0-19 points), 3 of the 4 questions utilize a range of 0-5 with 0 indicating the symptom is never experienced and 5 indicating the symptom is almost always experienced. The fourth question utilizes a range of 0-4 with 0 indicating the symptom is never experienced and 4 indicating the symptom is usually experienced. For the ICPI (score range: 0-16 points), all four questions utilize a range of 0-4 with 0 indicating it is no problem and 4 indicating it is a big problem.

SECONDARY OUTCOMES:
Complication rates between different hydrodistention parameters (pressure, number of distention, and duration of distention) | up to 30 days (after hydrodistention)
  These include bladder rupture, urinary tract infection/sepsis, prolonged retention, unplanned readmissions within 30 days.
Changes in the genitourinary pain index (GUPI) from baseline to 1- month | baseline to 1- month
  The GUPI questionnaire (score range: 0 - 45) contains nine overarching items related to urinary symptoms, pain, and impact on quality of life. A higher score denoting worse symptoms.
Changes in the genitourinary pain index (GUPI) from baseline to 1-week | baseline to 1-week
  The GUPI questionnaire (score range: 0 - 45) contains nine overarching items related to urinary symptoms, pain, and impact on quality of life. A higher score denoting worse symptoms.
Changes in the genitourinary pain index (GUPI) baseline to 3-months | baseline to 3-months
  The GUPI questionnaire (score range: 0 - 45) contains nine overarching items related to urinary symptoms, pain, and impact on quality of life. A higher score denoting worse symptoms.
Changes in the interstitial cystitis symptom index (ICSI) from baseline to 1-week | baseline to 1-week
  The O'Leary-Sant questionnaire is composed of the Interstitial Cystitis Symptom Index (ICSI) and Problem Index (ICPI) which contains four questions related to urinary and pain symptoms. For the ICSI (score range: 0-19 points), 3 of the 4 questions utilize a range of 0-5 with 0 indicating the symptom is never experienced and 5 indicating the symptom is almost always experienced. The fourth question utilizes a range of 0-4 with 0 indicating the symptom is never experienced and 4 indicating the symptom is usually experienced. For the ICPI (score range: 0-16 points), all four questions utilize a range of 0-4 with 0 indicating it is no problem and 4 indicating it is a big problem.
Changes in the interstitial cystitis symptom index (ICSI) from baseline to 3-months | baseline to 3-months
  The O'Leary-Sant questionnaire is composed of the Interstitial Cystitis Symptom Index (ICSI) and Problem Index (ICPI) which contains four questions related to urinary and pain symptoms. For the ICSI (score range: 0-19 points), 3 of the 4 questions utilize a range of 0-5 with 0 indicating the symptom is never experienced and 5 indicating the symptom is almost always experienced. The fourth question utilizes a range of 0-4 with 0 indicating the symptom is never experienced and 4 indicating the symptom is usually experienced. For the ICPI (score range: 0-16 points), all four questions utilize a range of 0-4 with 0 indicating it is no problem and 4 indicating it is a big problem.
Time spent in the post-anesthesia care unit (minutes) | After procedure (approximate time frame is 60 minutes)
Number of morphine milligram equivalents (MME) given in the post-anesthesia care unit | After procedure (approximate time frame is 1 hour)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No